CLINICAL TRIAL: NCT01682447
Title: Pulmonary Rehabilitation: Effects on Cognitive Functioning, Mood, Anxiety, and Quality of Life in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Pulmonary Rehabilitation: Effects on Cognitive Functioning, Mood, Anxiety, and Quality of Life in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tilburg University (Other)
Collaborators: Revant Schoondonck Center for Pulmonary Rehabilitation Breda (Unknown); Revant Innovation foundation (Unknown); Fonds NutsOhra (Other)
Responsible Party: Principal Investigator, Margriet M. Sitskoorn, Professor, PhD, Tilburg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NL33713.008.10
Record Dates: First submitted 2012-07-16; First posted 2012-09-11 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Chronic Obstructive Pulmonary Disease COPD
Keywords: COPD; Cognitive Dysfunction; Pulmonary Rehabilitation; Quality of life; Cognitive rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extensive Pulmonary Rehabilitation (ERP) (Experimental): Participants in this group are measured on primary and secondary outcome measures before and after a 12 week extensive pulmonary rehabilitation program.
  Interventions: Other: Extensive Pulmonary Rehabilitation Program
- Waiting List Control group (No Intervention): Participants in the waiting list control group are measured on primary and secondary outcome measures before and after waiting time for the extensive pulmonary rehabilitation program and start with this program after the second moment of measurement.

INTERVENTIONS:
Other: Extensive Pulmonary Rehabilitation Program — Fulltime pulmonary rehabilitation program. Duration: 12 weeks
  Arms: Extensive Pulmonary Rehabilitation (ERP)

SUMMARY:
The purpose of this project is to investigate whether a 12-week, fulltime pulmonary rehabilitation program can enhance cognitive functioning, mood, anxiety, and quality of life in patients with Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* COPD
* Referral to the Extensive Pulmonary Rehabilitation Program

Exclusion Criteria:

* Unfinished primary school
* Referral to the Compact Pulmonary Rehabilitation Program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in Objective Cognitive functioning | In the experimental group, this measure is assessed in the first and last week of rehabilitation with an average time frame of 11 weeks. In the Control group, this measure is assessed before and after waiting time with an average time frame of 5 weeks.
  CNS-Vital Signs, computerized neuropsychological assessment WMS - Verbal Paired Associates Direct Recall Word fluency-category (GIT): animals & profession Letter fluency: D-A-T Purdue Pegboard
Change in Mood and Anxiety | In the experimental group, this measure is assessed in the first and last week of rehabilitation with an average time frame of 11 weeks. In the Control group, this measure is assessed before and after waiting time with an average time frame of 5 weeks.
  Hospital Anxiety and Depression Scale (HADS)
  Symptom Checklist 90 - Revised (SCL-90-R), subscales Anxiety, Depression, Agoraphobia
Change in Quality of Life | In the experimental group, this measure is assessed in the first and last week of rehabilitation with an average time frame of 11 weeks. In the Control group, this measure is assessed before and after waiting time with an average time frame of 5 weeks.
  Saint George Respiratory Questionnaire (SGRQ)
  SF-36 Health Survey
Change in 6 Minute Walking distance Test(6-MWT) | In the experimental group, this measure is assessed in the first and last week of rehabilitation with an average time frame of 11 weeks. In the Control group, this measure is assessed before and after waiting time with an average time frame of 5 weeks.
  6 Minute Walking distance Test (6-MWT)
Change in Subjective Cognitive Functioning | In the experimental group, this measure is assessed in the first and last week of rehabilitation with an average time frame of 11 weeks. In the Control group, this measure is assessed before and after waiting time with an average time frame of 5 weeks.
  Cognitive Failures Questionnaire (CFQ)

SECONDARY OUTCOMES:
Adherence to pulmonary rehabilitation | These data are collected during the total period of pulmonary rehabilitation, which has a time frame of 12 weeks.
  Percentage of attendance of treatment session is collected from patients medical records.
  Adherence to pulmonary rehabilitation is specified as the percentage of the prescribed treatment sessions that patients actually attend. Adherence is further specified in the following categories: disease, motivation, other.
  We use this measure to explore the predictors (e.g., age, education, cognitive functioning) of adherence to pulmonary rehabilitation.
Change in Fatigue | In the experimental group, this measure is assessed in the first and last week of rehabilitation with an average time frame of 11 weeks. In the Control group, this measure is assessed before and after waiting time with an average time frame of 5 weeks.
  Chronic Respiratory Questionnaire (CRQ), subscale fatigue
Dropout from pulmonary rehabilitation | From the moment of randomization untill the moment of dropout from pulmonary rehabilitation, assessed up to 1 year after randomization.
  Dropout can be specified as the percentage of patients who, though eligible, do not start pulmonary rehabilitation or patients who do not finish pulmonary rehabilitation. Dropout is further specified in the following categories: death, disease, motivation, practical (e.g. move).
  We use this measure to explore the predictors (e.g., age, education, cognitive functioning) of dropout from pulmonary rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Margriet M. Sitskoorn, PhD., Principal Investigator — Tilburg University; Jan-Willem Meijer, MD., PhD., Study Chair — Revant Revalidatiecentrum Breda; Dirk Van Ranst, MD., Study Chair — Revant Revalidatiecentrum Breda; Carlijn A.M. Campman, MSc., Study Chair — Tilburg University
Locations (1):
- Revant Schoondonck Center for Pulmonary Rehabilitation, Breda, Netherlands